CLINICAL TRIAL: NCT00377923
Title: Endometrial Effects of Daily Progesterone s.c. 25 and 50 Mg Aqueous Formulation to Female Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05A/Prg05
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Last update posted 2006-09-20 (Estimated); Status verified 2006-09

CONDITIONS: Healthy
Keywords: pharmacodynamic and pharmacokinetic study; Progesterone; healthy volunteers; Endometrial decidualisation
MeSH Terms: interventions — Progesterone

INTERVENTIONS:
Drug: Progesterone

SUMMARY:
This is a multiple dose, observer blind, randomised, parallel groups pharmacodynamic and pharmacokinetic study to assess the endometrial effects (predecidual changes) of a new aqueous progesterone formulation administered s.c. at the dose of 25 and 50 mg/day.

DETAILED DESCRIPTION:
This study is designed in order to assess the efficacy of the investigational product (Progesterone acqueous s.c. formulation) when it is administered at the dose of 25 and 50 mg. The induced predecidual changes will be evaluated through endometrial bioptic samplings, performed on day 11 and will be compared between the two treatment groups.

The pharmacokinetic evaluation was designed according to internationally recognised guidelines for PK studies.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 19</=BMI</=25 kg/m2;
* Proper estrogen priming; absence of progesterone exposure prior to exogenous progesterone administration;
* normal pelvic ultrasound;
* absence of active follicular growth following initiation of E2 treatment;
* Complete suppression of ovarian function;
* Vital signs: SBP 100-139 mmHg, DBP 50-89, HR 50-90 bpm;
* Full comprehension of the nature and purpose of the study and possible risks and side effects;
* signed written informed consent prior to inclusion in the study

Exclusion Criteria:

* pregnant or lactating women;
* ECG: clinically relevant abnormalities;
* clinical relevant abnormal physical findings which could interfere with the objectives of the study;
* clinical relevant abnormal laboratory values indicative of physical illness, ascertained or presumptive hypersensitivity to the active principle and/or formulations' ingredients;
* history of anaphylaxis to drugs or allergic reactions in general, which the Investigator considers may affect the outcome of the study;
* history of uterine pathologies (fibroids, polyps, adenomyosis, etc), history of dysfunctional bleeding, relevant history of renal, hepatic, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases, history of neoplasias (genital apparatus, breast, liver or hormone-dependent cancer) severe liver failure, acute or chronic liver dysfunction, cholestatic jaundice, hypertension, thrombo-phlebitis, thrombo-embolism, cerebro-vascular insult or severe depression; medication, including OTC, during 2 weeks before the start of the study;
* participation in the evaluation of any drug within 1 month prior to the start of the study;
* blood donations during the 1 month prior to this study;
* history of drug, alcohol [>1 drink/day defined according to USDA Dietary Guidelines 2005 (18)] caffeine (>5 cups/ day of coffee or tea) or tobacco abuse (≥10 cigarettes/day);
* Abnormal diets (<1600 or >3500 kcal/day) or substantial changes in eating habits within the past 4 weeks.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24
Dates: Start 2005-08; Study Completion 2006-03

PRIMARY OUTCOMES:
partial and full predecidual changes in endometrial samples on the 11th day of exposure to the IMP compared to the findings on the 11th day after ovulation in the menstrual cycle, according to Noyes criteria

SECONDARY OUTCOMES:
PK profile of progesterone at the steady-state following the 25 or 50 mg/day of progesterone s.c. at the time of endometrial biopsy, local tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Markus Müller, Prof, Principal Investigator — Department of Clinical Pharmacology, AKH, Vienna, Austria.

REFERENCES:
- [Background] de Ziegler D, Bouchard P. Understanding endometrial physiology and menstrual disorders in the 1990s. Curr Opin Obstet Gynecol. 1993 Jun;5(3):378-88. PMID 8329654
- [Background] de Ziegler D, Bergeron C, Cornel C, Medalie DA, Massai MR, Milgrom E, Frydman R, Bouchard P. Effects of luteal estradiol on the secretory transformation of human endometrium and plasma gonadotropins. J Clin Endocrinol Metab. 1992 Feb;74(2):322-31. doi: 10.1210/jcem.74.2.1730810.
- [Background] NOYES RW, HAMAN JO. Accuracy of endometrial dating; correlation of endometrial dating with basal body temperature and menses. Fertil Steril. 1953 Nov-Dec;4(6):504-17. doi: 10.1016/s0015-0282(16)31446-7. No abstract available. PMID 13107761
- [Background] Noyes RW, Hertig AT, Rock J. Dating the endometrial biopsy. Am J Obstet Gynecol. 1975 May;122(2):262-3. doi: 10.1016/s0002-9378(16)33500-1. No abstract available. PMID 1155504
- [Background] Soliman S, Daya S, Collins J, Hughes EG. The role of luteal phase support in infertility treatment: a meta-analysis of randomized trials. Fertil Steril. 1994 Jun;61(6):1068-76. doi: 10.1016/s0015-0282(16)56758-2. PMID 8194619
- [Background] Pritts EA, Atwood AK. Luteal phase support in infertility treatment: a meta-analysis of the randomized trials. Hum Reprod. 2002 Sep;17(9):2287-99. doi: 10.1093/humrep/17.9.2287. PMID 12202415
- [Background] Bourgain C, Smitz J, Devroey P. Meta-analysis on luteal phase support. Hum Reprod. 2003 Mar;18(3):656; author reply 656-7. doi: 10.1093/humrep/deg098. No abstract available. PMID 12615845
- [Background] Daya S, Gunby J. Luteal phase support in assisted reproduction cycles. Cochrane Database Syst Rev. 2004;(3):CD004830. doi: 10.1002/14651858.CD004830. PMID 15266541
- [Background] de Ziegler D, Cornel C, Bergeron C, Hazout A, Bouchard P, Frydman R. Controlled preparation of the endometrium with exogenous estradiol and progesterone in women having functioning ovaries. Fertil Steril. 1991 Nov;56(5):851-5. doi: 10.1016/s0015-0282(16)54654-8. PMID 1936317
- [Background] Lelaidier C, de Ziegler D, Gaetano J, Hazout A, Fernandez H, Frydman R. Controlled preparation of the endometrium with exogenous oestradiol and progesterone: a novel regimen not using a gonadotrophin-releasing hormone agonist. Hum Reprod. 1992 Nov;7(10):1353-6. doi: 10.1093/oxfordjournals.humrep.a137572. PMID 1291558
- [Background] Fanchin R, De Ziegler D, Bergeron C, Righini C, Torrisi C, Frydman R. Transvaginal administration of progesterone. Obstet Gynecol. 1997 Sep;90(3):396-401. doi: 10.1016/s0029-7844(97)00270-6. PMID 9277651
- [Background] Gibbons WE, Toner JP, Hamacher P, Kolm P. Experience with a novel vaginal progesterone preparation in a donor oocyte program. Fertil Steril. 1998 Jan;69(1):96-101. doi: 10.1016/s0015-0282(97)00457-3. PMID 9457941
- [Background] Jobanputra K, Toner JP, Denoncourt R, Gibbons WE. Crinone 8% (90 mg) given once daily for progesterone replacement therapy in donor egg cycles. Fertil Steril. 1999 Dec;72(6):980-4. doi: 10.1016/s0015-0282(99)00390-8. PMID 10593367
- [Background] Damario MA, Barmat L, Liu HC, Davis OK, Rosenwaks Z. Dual suppression with oral contraceptives and gonadotrophin releasing-hormone agonists improves in-vitro fertilization outcome in high responder patients. Hum Reprod. 1997 Nov;12(11):2359-65. doi: 10.1093/humrep/12.11.2359. PMID 9436663
- [Background] de Ziegler D, Fanchin R. Progesterone and progestins: applications in gynecology. Steroids. 2000 Oct-Nov;65(10-11):671-9. doi: 10.1016/s0039-128x(00)00123-9. PMID 11108875
- [Derived] de Ziegler D, Sator M, Binelli D, Leuratti C, Cometti B, Bourgain C, Fu YS, Garhofer G. A randomized trial comparing the endometrial effects of daily subcutaneous administration of 25 mg and 50 mg progesterone in aqueous preparation. Fertil Steril. 2013 Sep;100(3):860-6. doi: 10.1016/j.fertnstert.2013.05.029. Epub 2013 Jun 24. PMID 23806850